CLINICAL TRIAL: NCT01305876
Title: Yoga in an Urban School for Children With Emotional Behavioral Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Naomi Steiner, Tufts Medical Center / Tufts University
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: 8756
Record Dates: First submitted 2011-02-18; First posted 2011-03-01 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-02

CONDITIONS: Emotional Behavioral Disorders
Keywords: yoga; emotional behavioral disorder; intervention; school; meditation; focus: yoga intervention in students with emotional behavioral disorders in an urban school

ARMS (1):
- one group with yoga intervention (Experimental): one group with yoga intervention
  Interventions: Behavioral: yoga intervention

INTERVENTIONS:
Behavioral: yoga intervention — yoga session 2 x week over 3-1/2 months

SUMMARY:
Yoga is becoming a part of therapies for children with emotional behavioral disorders. The goal is to examine the feasibility and efficacy of yoga sessions for children with emotional behavioral disorders at an urban elementary school.

DETAILED DESCRIPTION:
Participants: children in 4th and 5th grade at an urban elementary school, identified by the special education director and the teaching staff, as having emotional behavioral disorders including anxiety, depression, aggression, conduct disorder, hyperactivity and attention difficulties. These grades have a combined student population of 160 students. Enrolled over two years.

Inclusion/Exclusion criteria:

Eligible if identified by the teaching staff or special education director as having an emotional behavioral disorder. Exclusion criteria: inability to comprehend English sufficiently to complete written assessments and follow the yoga intervention.

Pre- and post-intervention assessments (teachers)

1. Behavior Assessment Scale for Children (BASC).
2. The Swanson, Kotkin, Agler, M-Flynn & Pelham Rating Scale (SKAMP)

ELIGIBILITY:
Inclusion Criteria:

* identified by the teaching staff or special education director as having an emotional -behavioral disorder

Exclusion Criteria:

* inability to comprehendread in English sufficiently to complete written assessments and follow the yoga interventionintervention protocols

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2008-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Behavior Assessment Scale for Children (BASC). | 1 year. The classroom teachers filled out the BASC pre- and post-intervention on each participant. This took place June 2009, after the yoga intervention took place. Has been completed
  The BASC was chosen to track the effect of the yoga intervention on classroom behavior. The BASC is a tool tht is frequently used within the school setting to track classroom behavior and overall wellbeing of students. The BASC has been shown to have adequate reliability and validity based on concurrence with similar scales (Reynolds & Kamphaus, 1992). Subscales include anxiety, aggression, attention problems, hyperactivity, conduct problems, depression, withdrawal and social skills.
The Swanson, Kotkin, Agler, M-Flynn & Pelham Rating Scale (SKAMP) | One year. The teachers filled out the SKAMP pre- and post-intervetnion to assess participants focus in class. This took place June 2009, after the yoga interveniton. Has been completed.
  The SKAMP was used for teachers to assess classroom attention. The SKAMP is a validated teacher observation assessment rating scale composed of 10 items, designed to describe classroom behavior and attention (Gansle et al., 2004; Sharon, Wigal, & Wigal, 2006).The SKAMP is used to monitor interventions and has been shown to be sensitive to change (McBurnett, Swanson, Pfiffner, & Tam, 1997).

SECONDARY OUTCOMES:
The Swanson, Kotkin, Agler, M-Flynn & Pelham Rating Scale (SKAMP) | The classroom teachers filled out the SKAMP pre- and post-intervention
  The SKAMP was filled out by classroom teachers to assess students' ability to pay attention in class. It is a validated teacher observation assessment rating scale composed of 10 items, designed to describe classroom behavior and attention (Gansle et al., 2004; Sharon, Wigal, & Wigal, 2006).The SKAMP is used to monitor interventions and has been shown to be sensitive to change (McBurnett, Swanson, Pfiffner, & Tam, 1997).

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts Medical Center / Tufts University, Boston, Massachusetts, United States